CLINICAL TRIAL: NCT00371111
Title: To Compare Therapeutic Effect of Intravitreal Bevacizumab and Triamcinolone in Resistant Uveitic Cystoid Macular Edema
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8524
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Resistant Cystoid Macular Edema
Keywords: Resistant uveitic cystoid macular edema; intravitreal triamcinolone; intravitreal bevacizumab

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator): Intravitreal injection of Triamcinolone
  Interventions: Drug: Intravitreal injection of Triamcinolone
- 2 (Active Comparator): Intravitreal injection of Avastin
  Interventions: Drug: Intravitreal injection of Avastin

INTERVENTIONS:
Drug: Intravitreal injection of Triamcinolone — 4 mg of Triamcinolone
  Arms: 1
Drug: Intravitreal injection of Avastin — Injection of 1.25 mg of Avastin and
  Arms: 2

SUMMARY:
Cystoid macular edema (CME) is one of the common causes of vision loss in patients with UveitiS .Triamcinolone has been effectively used in reducing CME and improving the vision. Also there are some documents which recommend Bevacizumab(avastin) could reduce macular edema. This study compare intravitreous injection of triamcinolone and avastin in patients with resistant uveitic cystoid macular edema.

DETAILED DESCRIPTION:
This study compare intravitreous injection of triamcinolone and avastin in patients with resistant uveitic cystoid macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Uveitic CME
* Uveitic CME refractory to routine treatment
* Vision better than 5/200 and worse than 20/50

Exclusion Criteria:

* Mono- Ocular patients
* History of vitrectomy
* Glaucoma or ocular hypertension
* History of other retinal disease that can cause macular edema
* Pregnancy
* Significant media opacity
* Vision better than 20/50

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Resorbed CME in OCT | every 3 month
Resorbed CME in clinical examination | Every 3 month

SECONDARY OUTCOMES:
need to retreatment | when ever needed

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Soheilian, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Masoud Soheilian , MD, Tehran, Tehran Province, Iran